CLINICAL TRIAL: NCT00457574
Title: A Single-Center, Open-Label, Phase I Study of Single-Agent GMX1777 Administered as a 24-Hour Infusion Every 3 Weeks to Patients With Refractory Solid Tumors or Lymphomas
Brief Title: Safety and Efficacy of GMX1777 in the Treatment of Refractory Solid Tumors or Lymphomas
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated prematurely due to financial constraints.
Sponsor: Gemin X (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM301
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Solid Tumors and Lymphomas
MeSH Terms: conditions — Lymphoma | interventions — 1-(2-(2-(2-(2-methoxyethoxy)ethoxy)ethoxy)ethoxycarbonyloxymethyl)-4-(N'-cyano-N''-(6-(4-chlorophenoxy)hexyl)-N-guanidino)pyridinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GMX1777

SUMMARY:
GMX1777 is a water-soluble, intravenously-administered prodrug of GMX1778. GMX1777 is rapidly converted to GMX1778 in vivo. GMX1778 has potent anti-tumor activity against a variety of cell lines and models from different tumor origins.

DETAILED DESCRIPTION:
This is a single-center, open-label, Phase I study of single-agent GMX1777 administered every 3 weeks to patients with CLL, MM, refractory solid tumors or lymphomas. No investigational or commercial agents or therapies other than those described may be administered with the intent to treat the patient's malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed solid tumor or lymphoma
* No limitations on allowable type and amount of prior therapy.
* Patients must have a life expectancy of greater than 8 weeks
* Patients must have normal organ and marrow function
* Patients must be willing to submit blood sampling for planned PK analysis
* Patients must have the ability to understand and willingness to sign a written informed consent form

Exclusion Criteria:

* No other agents or therapies administered with the intent to treat malignancy
* Patients with prior exposure to GMX1777 or GMX1778
* Uncontrolled, intercurrent illness
* Pregnant women and women who are breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2009-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Determine the recommended Phase II dose; Characterize the dose-limiting toxicities; Determine the pharmacokinetic parameters | 52 weeks

SECONDARY OUTCOMES:
Describe observed tumor responses | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Berger, MD, Study Director — Gemin X, Inc.